CLINICAL TRIAL: NCT05871723
Title: The Relationship of Multifidus and Gastrocnemius Muscle Thickness With Postural Stability in Patients With Stroke
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uskudar State Hospital (Other Government)
Collaborators: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Principal Investigator, Uskudar State Hospital
Other Study IDs: SVOposture1
Record Dates: First submitted 2023-05-08; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Stroke; Postural; Defect; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke Patients: Patients diagnosed with stroke.
  Interventions: Other: Measurement of multifidus and gastrocnemius muscle thickness with Ultrasound; Other: Berg Balance Scale

INTERVENTIONS:
Other: Measurement of multifidus and gastrocnemius muscle thickness with Ultrasound — o measure multifidus and gastrocnemius muscle thickness using ultrasound imaging, the following steps are typically followed. First, the patient is positioned appropriately to allow access to the muscles to be imaged. For example, the patient may lie prone for imaging of the lumbar multifidus or sit with the leg extended for imaging of the gastrocnemius. Next, a trained clinician or technician places an ultrasound probe on the skin over the target muscle and adjusts the settings on the ultrasound machine to optimize the image quality. The probe is then moved around to obtain different views of the muscle, and the images are stored for later analysis. To measure muscle thickness, the clinician or technician identifies the muscle fascia on the ultrasound image and measures the distance between the fascia and the underlying bone or tissue. This measurement provides an estimate of the muscle thickness.
Other: Berg Balance Scale — The Berg Balance Scale is a clinical assessment tool used to measure an individual's ability to maintain balance during various functional tasks. The test includes 14 items, such as standing unsupported, reaching forward, turning, and standing on one leg. Each item is scored on a 5-point scale, ranging from 0 (unable to perform the task) to 4 (able to perform the task independently and safely). The scores for each item are summed to provide a total score, with a maximum possible score of 56. The Berg Balance Scale is commonly used in clinical and research settings to assess balance impairment and monitor changes in balance over time, particularly in individuals with neurological conditions such as stroke. The test has good reliability and validity and is considered a gold standard for assessing balance in these populations.

SUMMARY:
This study aims to investigate the relationship between multifidus and gastrocnemius muscle thickness with postural stability in patients with stroke.

DETAILED DESCRIPTION:
Multifidus and gastrocnemius muscle thickness will be measured using ultrasound imaging. Postural stability will be assessed using the Berg Balance Scale, a clinical balance test that assesses an individual's ability to maintain balance during various functional tasks. The Berg Balance Scale includes 14 items, such as standing unsupported, reaching forward, turning, and standing on one leg. The Berg Balance Scale is a widely used clinical balance test that has good reliability and validity in stroke patients. Data will be analyzed using appropriate statistical methods, including correlation and regression analysis, to investigate the relationship between the multifidus and gastrocnemius muscle thickness and postural stability.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stroke: Patients who have a confirmed diagnosis of stroke based on medical history, clinical examination, and diagnostic imaging.
* Time since stroke onset: The trial may include patients who are at least 6 months post-stroke onset.
* Ability to understand instructions: Patients who are able to understand and follow instructions provided for the study procedures.
* Ability to provide informed consent: Patients who are able to provide informed consent or have a legal representative who can provide informed consent on their behalf.

Exclusion Criteria:

* Cognitive impairment: Patients who have significant cognitive impairment that may affect their ability to follow instructions or participate in the study procedures.
* Severe motor deficits: Patients with severe motor deficits that may limit their ability to perform the study procedures.
* Other medical conditions: Patients with other medical conditions or comorbidities that may affect muscle thickness or postural stability, such as Parkinson's disease, multiple sclerosis, or severe osteoarthritis.
* Inability to tolerate testing: Patients who are unable to tolerate the testing procedures, such as the Berg Balance Scale or ultrasound imaging.
* Implanted devices: Patients with implanted devices, such as pacemakers, that may be affected by the ultrasound imaging.
* Not giving consent.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stroke patients who gave consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Relationship between multifidus thickness and postural stability | 1 day
  he relationship between multifidus muscle thickness measured by ultrasound in cm and results of berg scale will be measured statistically by calculating correlation coefficients.
  The Berg Balance Scale is a widely used clinical assessment tool designed to measure balance and stability in individuals who may have balance impairments due to various conditions such as stroke, Parkinson's disease, or multiple sclerosis. It consists of a series of 14 balance-related tasks that assess various aspects of balance, including sitting balance, standing balance, and dynamic balance.
  Each task is scored on a 5-point scale ranging from 0 to 4, with higher scores indicating better balance performance. The tasks involve different movements and challenges, such as maintaining sitting balance without arm support, standing up from a seated position, reaching forward while standing, turning around, and maintaining balance in different standing positions.
Relationship between gastrocnemius muscle thickness and postural stability | 1 day
  The relationship between gastrocnemius muscle thickness measured by ultrasound in cm and results of berg scale will be measured statistically by calculating correlation coefficients.
  The Berg Balance Scale is a widely used clinical assessment tool designed to measure balance and stability in individuals who may have balance impairments due to various conditions such as stroke, Parkinson's disease, or multiple sclerosis. It consists of a series of 14 balance-related tasks that assess various aspects of balance, including sitting balance, standing balance, and dynamic balance.
  Each task is scored on a 5-point scale ranging from 0 to 4, with higher scores indicating better balance performance. The tasks involve different movements and challenges, such as maintaining sitting balance without arm support, standing up from a seated position, reaching forward while standing, turning around, and maintaining balance in different standing positions.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa H Temel, M.D., Principal Investigator — Uskudar State Hospital

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be shared upon reasonable request by the corresponding author.